CLINICAL TRIAL: NCT01437436
Title: The Effect of Obesity on Ventilation Tube Insertion
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Soonchunhyang University Hospital (Other)
Responsible Party: Principal Investigator, Park Moo Kyun, Assistant professor, Soonchunhyang University Hospital
Other Study IDs: SCHBC-11501
Record Dates: First submitted 2011-09-19; First posted 2011-09-20 (Estimated); Last update posted 2011-09-23 (Estimated); Status verified 2011-09

CONDITIONS: Otitis Media; Obesity
Keywords: otitis media; obesity; ventilation tube
MeSH Terms: conditions — Otitis Media; Obesity | interventions — Middle Ear Ventilation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- obesity: otitis media patient with obesity
  Interventions: Procedure: ventilation tube
- non obesity: otitis media patient with non obesity
  Interventions: Procedure: ventilation tube

INTERVENTIONS:
Procedure: ventilation tube — ventilation tube insertion

SUMMARY:
Obesity is associated with increased risk of surgical complications. Ventilation tube insertion is one of the most frequent surgical procedures performed on children. However, the impact of obesity on surgical results or surgical related complication following ventilation tube insertion remains poorly understood. The aim of this study was to investigate the effect of obesity on the surgical results of ventilation tube insertion for otitis media with effusion (OME) in pediatric patients.

DETAILED DESCRIPTION:
OME was diagnosed by the presence of fluid in the middle ear on otoscopy or tympanometry according to clinical practice guidelines . The diagnostic findings of pneumatic otoscopy and otomicroscopy include the tympanic membrane dullness, impaired mobility, and an air-fluid level or bubble. In addition, the type B or C tympanogram was considered positive for OME.

Indication for ventilation tub insertion includes history of OME lasting 3 months or longer, structural damage to tympanic membrane or middle ear and risk for speech, language learning difficulties. Adenoidectomy is also performed when adenoid hypertrophy is founded during preoperative assessment.

Body weight and height were measured before ventilation tube insertion at hospital. Body mass index (BMI) was calculated using the formula weight/ height2 (Kg/m2).

ELIGIBILITY:
Inclusion Criteria:

* Children aged 2-15 years with a diagnosis of OME who underwent ventilation tube insertion

Exclusion Criteria:

* Children with a previous history of ventilation tube insertion
* Use of ventilation tubes other than Paparella type I
* Head and neck anomalies
* Chronic or systemic disease

Ages: 2 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Residents of bucheon city in South Korea
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2010-10; Primary Completion 2012-06 (Estimated); Study Completion 2012-06 (Estimated)